CLINICAL TRIAL: NCT04717063
Title: Clinical Efficacy of Single-Use of Peroxyl Mouthwash for Reducing Bacteria in Saliva and Bioaerosol Contamination Phase 2
Brief Title: Clinical Efficacy of Single-Use of Peroxyl Mouthwash for Reducing Bacteria Saliva and Bioaerosol Contamination Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2020-08-BAC-HP-CA-BGS2
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Mouthwash; Saliva; Bioaerosol; Bacteria; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to receive one of the two possible study products
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peroxyl (Active Comparator): Drug: Peroxyl Mouthwash Mouthwash
  Other Names:
  • 1.5% HP
  Interventions: Drug: Peroxyl Oral Product
- placebo mouthwash (Placebo Comparator): Drug: Placebo Mouthwash Mouthwash
  Other Names:
  • 0.0% HP Mouthwash
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peroxyl Oral Product — mouth wash
  Other Names: Peroxyl Mouth wash
  Arms: Peroxyl
Drug: Placebo — placebo mouth wash
  Arms: placebo mouthwash

SUMMARY:
To evaluate the antibacterial efficacy of a commercial mouthwash containing 1.5% hydrogen peroxide in reducing the levels of bacteria in bioaerosols generated by dental prophylaxis.

DETAILED DESCRIPTION:
Following a washout period, subjects will return to the clinical site. A baseline microbial sample will be collected from the operatory's atmosphere for 30 min. prior to the study subject appointment by placing blood agar plates on a support board attached to the bracket chair tray. Upon completion of a half-mouth (e.g. right side) dental prophylaxis, each study subject will be instructed to rinse for one minute with 10 ml of one of the two mouthwash solutions (1.5% hydrogen peroxide or 0.0% hydrogen peroxide) and to expectorate all remaining liquid. Next, the dental prophylaxis will be completed on the other side of the mouth. Bioaerosol samples will be collected prior to and following rinsing on blood agar plates placed on a support board at a 50-degree angle to the participant's chest, on the participant's chest, and on the examiner's forehead. Plates will be closed and labeled. The plates will be transferred to the microbiology laboratory for analysis. All subjects will be followed for adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must meet ALL of the following criteria:

  * Subjects, ages 18-70, inclusive.
  * Availability for the duration of this clinical research study.
  * Good general health.
  * At least 20 natural teeth.
  * Gingivitis Index 1.0 (Löe-Silness).
  * Signed Informed Consent Form

Exclusion Criteria:

* Potential subjects must NOT HAVE ANY of the following conditions:

  * Symptoms consistent with COVID-19 or have tested positive.
  * Presence of orthodontic bands.
  * Tumor(s) of the soft or hard tissues of the oral cavity.
  * Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone) or peri-implantitis.
  * Five or more carious lesions requiring immediate restorative treatment.
  * Use of antibiotic one-month prior to entry into the study.
  * Participation in any other clinical study or test panel within the one month prior to entry into the study.
  * Dental prophylaxis during the past two weeks prior to baseline examinations.
  * History of allergies to oral care/personal care consumer products or their ingredients.
  * On any prescription medicines that might interfere with the study outcome.
  * An existing medical condition that prohibits not eating or drinking for periods up to 4 hours.
  * History of alcohol or drug abuse.
  * Self-reported pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
evaluate the antibacterial efficacy of mouthwash in reducing the levels of bacteria in bioaerosols generated by dental prophylaxis | 30 min
  baseline microbial sample will be collected from the operatory's atmosphere for 30 min. prior to the study subject appointment by placing blood agar plates on a support board attached to the bracket chair tray. Upon completion of a half-mouth (e.g. right side) dental prophylaxis, each study subject will be instructed to rinse for one minute with 10 ml of one of the two mouthwash solutions (1.5% hydrogen peroxide or 0.0% hydrogen peroxide) and to expectorate all remaining liquid. Next, the dental prophylaxis will be completed on the other side of the mouth. Bioaerosol samples will be collected prior to and following rinsing on blood agar plates placed on a support board at a 50-degree angle to the participant's chest, on the participant's chest, and on the examiner's forehead. Plates will be closed and labeled. The plates will be transferred to the microbiology laboratory for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, DDS MSD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No